CLINICAL TRIAL: NCT06446206
Title: Adebrelimab Plus Chemotherapy and Bevacizumab Induction Therapy Followed by Maintenance Therapy With Adebrelimab Plus Fluzoparib and Bevacizumab in Platinum-Sensitive Relapsed Ovarian Cancer (CHANGCHUN): A Single-Arm, Exploratory Study
Brief Title: Adebrelimab Plus Chemotherapy, Bevacizumab and Fluzoparib in Platinum-Sensitive Relapsed Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ziling Liu, Principal Investigator, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-HS-022
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Platinum-sensitive Relapsed Ovarian Cancer
MeSH Terms: interventions — Paclitaxel; Carboplatin; Bevacizumab; fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Drug: Adebrelimab, paclitaxel, carboplatin, bevacizumab, fluzoparib

INTERVENTIONS:
Drug: Adebrelimab, paclitaxel, carboplatin, bevacizumab, fluzoparib — Adebrelimab plus paclitaxel, carboplatin and bevacizumab induction therapy followed by maintenance therapy with adebrelimab plus fluzoparib and bevacizumab.

SUMMARY:
The investigators explore the efficacy and safety of adebrelimab (PD-L1 inhibitor) plus chemotherapy and bevacizumab induction therapy followed by maintenance therapy with adebrelimab plus fluzoparib (PARP inhibitor)and bevacizumab in platinum-sensitive relapsed ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study after full informed consent and signed a written informed consent form;
2. Aged 18-75 years old;
3. Pathologically confirmed ovarian epithelial cancer, epithelial fallopian tube cancer, or primary peritoneal cancer;
4. International Federation of Gynecology and Obstetrics (FIGO) 2018 edition staging III-IV;
5. Having received no more than 2 prior lines of platinum-containing chemotherapy and ≥ 6 months between the time of last chemotherapy and tumor recurrence;
6. No more than 1 prior PARP inhibitor;
7. Negative for germline breast cancer susceptibility gene(BRCA) mutations;
8. At least 1 measurable lesion according to RECIST 1.1 evaluation criteria;
9. Patients with expected survival of ≥12 weeks;
10. Have an Eastern Cooperative Oncology Group(ECOG) Performance Status(PS) score of 0-1;
11. The patient has good organ function: without having received transfusions of blood products, granulocyte colony-stimulating factor, interleukin 11, thrombopoietin, or thrombopoietin receptor agonists within 14 days prior to the first receipt of therapeutic agents in this regimen：

    * Neutrophil count ≥1.5 x 10^9/L.
    * platelet count ≥ 80 × 10^9/ L.
    * hemoglobin ≥75 g/L.
    * albumin ≥30 g/L.
    * Albumin ≥30 g/L
    * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
    * Alanine amino transferase(ALT), Aspartate amino transferase(AST) ≤ 3 times ULN (without liver metastases) or ≤ 5 times ULN (if liver metastases occur)
    * Serum creatinine ≤1.5 times upper limit of normal (ULN)
    * Requirements for coagulation: international normalized ratio (INR) ≤1.5 times ULN, prothrombin time (PT) ≤1.5 times ULN, activated partial thromboplastin time (APTT) ≤1.5 times ULN.
    * Corrected serum electrolytes within normal range;
12. Women of childbearing potential must have had a negative pregnancy test (serum or urine) within 7 days prior to enrollment and be willing to use an appropriate method of contraception for the duration of the trial and for 8 weeks after the last administration of the test drug.

Exclusion Criteria:

1. Known hypersensitivity or severe allergic reactions to the study drug or any of its excipients;
2. Concurrent other incurable malignancies;
3. The presence of uncontrolled or symptomatic active central nervous system (CNS) metastases;
4. Pregnancy or confirmed by blood or urine Human Chorionic Gonadotropin(HCG) test or lactation, or subjects of childbearing potential who are unwilling or unable to use effective contraception (for both male and female subjects) until at least 6 months after the last trial treatment;
5. Difficult-to-control diabetes mellitus (defined as high fluctuations in blood glucose that interfere with the patient's life as well as frequent hypotension despite standard insulin therapy and frequent blood glucose monitoring);
6. Myocardial infarction, severe/unstable angina pectoris, New York Heart Association(NYHA) class 2 or greater cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmias and symptomatic congestive heart failure, uncontrolled hypertension of moderate or greater severity (Systolic Blood Pressure >160 mm Hg or Diastolic Blood Pressure >100 mm Hg) within 4 weeks prior to the first study dose, known coronary artery disease, congestive heart failure that does not meet the above criteria congestive heart failure or left ventricular ejection fraction <50% that meets the above criteria must be treated with an optimally stabilized medical regimen as determined by the treating physician and, if appropriate, in consultation with a cardiologist;
7. Patients with a history of neurologic autoimmune disease, or moderate to severe autoimmune disease, or high doses of immunosuppressive agents for symptom control
8. History of known allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
9. Receipt of any of the following medications or treatments prior to the first study drug treatment

   1. major surgery within 6 weeks (tissue biopsies and Peripherally Inserted Central Catheter or infusion port implantation via peripheral venous puncture for diagnostic purposes are permitted)
   2. Requires ongoing high-dose systemic corticosteroids (>10 mg/day prednisone or equivalent dose of other medications) or other systemic immunosuppressants (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, tacrolimus, cyclosporine, meclofenamic acid esters, anti-thymocyte globulin, and anti-tumor necrosis factor medications), and continues to be required after enrollment; [Note]: Topical skin, ocular, intra-articular, intranasal, and inhaled corticosteroids are permitted .
10. Serious infections within 90 days, such as severe pneumonia requiring hospitalization, bacteremia, and co-infections; active tuberculosis; [Note 1] Hepatitis B Surface Antigen Positive (HBsAg+) and/or Hepatitis B Core Antibody Positive (HBcAb+) patients will be required to undergo a Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) test, if the HBV DNA copy number <1000 cps/mL, or less than the lower limit of detectable value of the research center, can participate in this study and regulate the use of anti-hepatitis B virus medication; [Note 2] patients with hepatitis C antibody positive (HCV Ab+) need to undergo HCV RNA testing, and HCV RNA negative (defined as less than the lower limit of detectable value of the research center) can participate in this study;
11. Psychiatric disorders that interfere with informed consent and/or protocol adherence;
12. Other conditions that, in the judgment of the investigator, make participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
12-month progression-free survival rate | Twelve months after patients received their first antitumor drug therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | The radiological evaluations will be performed once at the end of every 2 cycles within 6 cycles and once every 4 cycles after Cycle 6(each cycle is 21 days).
Progression-free survival of CR/PR | The time from the first dose of investigational product to the first progression of disease (PD) in radiological evaluation or death for any reason (whichever comes first), assessed up to 2 years .
  Progress Free Survival (PFS) in patients with complete response (CR)/partial response (PR) after induction chemotherapy.
Progression-free survival of SD | The time from the first dose of investigational product to the first progression of disease (PD) in radiological evaluation or death for any reason (whichever comes first), assessed up to 2 years .
  Progress Free Survival (PFS) in patients with stable disease (SD) after induction chemotherapy.
Overall Survival（OS） | The time from the first dose of investigational product to the death for any reason, assessed up to 2 years.

OTHER OUTCOMES:
All grades adverse event (AE) | Through study completion, an average of 2 year.
  Classification per Common Terminology Criteria for Adverse Events (CTC-AE) version 5.0.
Serious adverse events | Through study completion, an average of 2 year.
  ≥ grade 3 per CTC-AE version 5.0.
Immune checkpoint inhibitor-related adverse events（irAEs） | Through study completion, an average of 2 year.

IPD SHARING:
Plan to Share IPD: Undecided